CLINICAL TRIAL: NCT04609176
Title: A Prospective, Non-randomized, Multicenter, Phase II Study of Camrelizumab (SHR-1210) and Apatinb Based Therapies for Unresectable Recurrent or Metastatic Alpha-fetoprotein (AFP)-Producing Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of Camrelizumab (SHR-1210) and Apatinb Based Therapies for Alpha-fetoprotein (AFP)-Producing Gastric Cancer or Gastroesophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-007
Record Dates: First submitted 2020-10-17; First posted 2020-10-30 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab+Apatinib+SOX (Experimental): Participants who have not received any previous therapy for their disease will receive Camrelizumab and Apatinib in combination with Oxaliplatin and S-1. Camrelizumab 200mg, day1; Apatinib 250mg qd p.o.;Oxaliplatin 130 mg/m2 day1; S-1 40-60 mg (calculated according to the body surface area) bid day1-14. 3 weeks for one cycle.
  Interventions: Drug: Camrelizumab plus Apatinib and SOX
- Camrelizumab+Apatinib (Experimental): Participants who have received at least one prior therapy for their advanced disease will receive Camrelizumab and Apatinib. Camrelizumab 200mg, day1; Apatinib 250mg qd p.o. 3 weeks for one cycle.
  Interventions: Drug: Camrelizumab plus Apatinib

INTERVENTIONS:
Drug: Camrelizumab plus Apatinib and SOX — Camrelizumab 200mg, day1; Apatinib 250mg qd p.o.;Oxaliplatin 130 mg/m2 day1; S-1 40-60 mg (calculated according to the body surface area) bid day1-14. 3 weeks for one cycle.
  Arms: Camrelizumab+Apatinib+SOX
Drug: Camrelizumab plus Apatinib — Camrelizumab 200mg, day1; Apatinib 250mg qd p.o. 3 weeks for one cycle.
  Arms: Camrelizumab+Apatinib

SUMMARY:
This is a study of Camrelizumab (SHR-1210) and Apatinb for unresectable Recurrent or metastatic alpha-fetoprotein (AFP)-producing gastric cancer or Gastroesophageal Junction Adenocarcinoma. Camrelizumab combined with Apatinib and standard chemotherapy will be given to treatment-naïve participants; Camrelizumab combined with Apatinib will also be evaluated in participants who have had ≥ 1 line of previous treatment. The primary endpoint is the Overall Response Rate (ORR).

DETAILED DESCRIPTION:
This study will have 2 cohorts. In Cohort 1, participants who have not received any previous therapy for their disease will receive Camrelizumab and Apatinib in combination with Oxaliplatin and S-1. In Cohort 2, participants who have received at least one prior therapy for their advanced disease will receive Camrelizumab and Apatinib. A Simon two-stage phase II design was used for the sample size Calculation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provided written informed consent to be subjects in this trial
2. Aged ≥18 years
3. Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
4. Has histologically-confirmed diagnosis of locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma
5. Clinical staging was performed according to enhanced CT/MRI examination (combined with endoscopic ultrasonography and diagnostic laparoscopic exploration if necessary). For patients with locally advanced or metastatic gastric/GEJ cancer in stage III-IV (AJCC 8 edition TNM stage) that could not be resected, the possibility of resectable was determined by MDT
6. For cohort 1, no prior systemic chemotherapy for the treatment of the participant's advanced or metastatic disease (treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as completed at least 6 months prior to the diagnosis of advanced or metastatic disease); for cohort 2, received and progressed on ≥1 prior systemic therapy for their advanced disease.
7. Have measurable disease as defined by RECIST 1.1 as determined by investigator assessment
8. Serum AFP > 2 upper limit of normal (ULN) or AFP positive by immunohistochemical staining methods
9. Adequate Organ Function Laboratory Values:

   Hemoglobin ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelets ≥80×109/L; AST and ALT ≤ 2.5 ULN or ≤ 5 ULN for subjects with liver metastases; Total bilirubin ≤1.5 ULN; Serum creatinine ≤1.5 ULN or measured or calculated creatinine clearance > 50ml/min; Albumin ≥ 30g/L;
10. No serious concomitant disease result in survival of less than 5 years
11. Patients capable of taking oral medication
12. Have good compliance and be able to follow the study protocol
13. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication and must be willing to use an adequate method of contraception for the course of the study through 90 days after the last dose of study medication. Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy
14. Agree to provide blood and/or tumor tissue sample deemed adequate for PD-L1 and other biomarker analysis.

Exclusion Criteria:

1. Is pregnant or breastfeeding
2. HER2 positive subjects will be excluded from cohort 1
3. Patients have recovered adverse events associated with pretreatment to Grade 1 or lower with CTCAE v5.0 excluding alopecia
4. Patients have an active malignancy (except for definitively treated basal cell carcinoma of the skin, or carcinoma-in-situ of the cervix) within the past 5 years
5. Active heart disease that is not well controlled, e.g. symptomatic coronary heart disease, New York Heart Association (NYHA) congestive heart failure of grade II or above, severe arrhythmias requiring drug intervention, myocardial infarction within the past 12 months, QTc ≥ 450ms for male, QTc ≥ 450ms for female, LVEF<50%
6. Genetic or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulation disorders, thrombocytopenia, etc.)
7. Patients with a history of gastrointestinal perforation, intra-abdominal abscess, or in-three-months ileus
8. Coagulation disorders (International normalized ratio, INR > 2.0 or Prothrombin time, PT > 16s)
9. Organ transplantation requires immunosuppressants, or who have received immunosuppressants/systemic corticosteroids therapy <14 days before first dose for an immunosuppression purpose (> 10mg/day prednisone or other equivalency drugs)
10. Patients have an active ulcer, serious non-healing wound, or bone fracture
11. Patients with hypertension that is difficult to control (systolic blood pressure ≥140 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents
12. Patients have a deficiency of dihydropyrimidine dehydrogenase (DPD) will be excluded from cohort 1
13. Have any contraindications for study treatment
14. Patients with a history of prior treatment with Apatinib or any anti-PD-1, anti-PD-L1 agent
15. Urinary protein is more than 2+ and 24-hour urine protein > 1.0g
16. Patients with active hepatitis B (HBsAg positive and HBV DNA≥500 IU/ml), hepatitis C (HCV antibodies positive and HCV RNA copies > ULN); with active infection requiring drug intervention
17. Patients with active symptoms or signs of interstitial lung disease
18. Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease
19. Patients were judged unsuitable as subjects of this trial by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) According to RECIST 1.1 based on investigator assessment | Up to approximately 24 months
  ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR according to RECIST 1.1 based on investigator assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) According to iRECIST 1.1 based on investigator assessment | Up to approximately 24 months
  ORR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR according to iRECIST 1.1 based on investigator assessment.
Disease Control Rate (DCR) According to RECIST 1.1 based on investigator assessment | Up to approximately 24 months
  DCR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR or SD according to RECIST 1.1 based on investigator assessment.
Duration of Response (DOR) According to RECIST 1.1 Based on investigator assessment | Up to approximately 24 months
  DOR was defined as the time from first documented evidence of CR or PR until disease progression (according to RECIST 1.1 )or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) According to RECIST 1.1 base on investigator assessment | Up to approximately 24 months
  PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) According to iRECIST 1.1 base on investigator assessment | Up to approximately 24 months
  DCR was defined as the percentage of the participants in the analysis population who had a confirmed CR or PR or SD according to iRECIST 1.1 based on investigator assessment.
Duration of Response (DOR) According to iRECIST 1.1 base on investigator assessment | Up to approximately 24 months
  DOR was defined as the time from first documented evidence of CR or PR until disease progression (according to iRECIST 1.1) or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) According to iRECIST 1.1 base on investigator assessment | Up to approximately 24 months
  PFS was defined as the time from randomization to the first documented disease progression per iRECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 24 months
  OS was defined as the time from randomization to death due to any cause.
Number of Participants Experiencing an Adverse Event (AE) | Up to approximately 27 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an adverse event. The number of participants who experienced an AE was reported for each arm according to the treatment received. The grade of AE will be assessed per CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China

REFERENCES:
- [Derived] Wang Y, Lu J, Chong X, Wang C, Chen X, Peng Z, Gu Y, Wang Y, Wang X, Li J, Gong J, Qi C, Yuan J, Lu Z, Lu M, Zhou J, Cao Y, Chen Y, Zhang C, Hou Z, Kou H, Shen L, Zhang X. PD-1 antibody camrelizumab plus apatinib and SOX as first-line treatment in patients with AFP-producing gastric or gastro-esophageal junction adenocarcinoma (CAP 06): a multi-center, single-arm, phase 2 trial. Signal Transduct Target Ther. 2025 Mar 14;10(1):100. doi: 10.1038/s41392-025-02193-z. PMID 40082418